CLINICAL TRIAL: NCT03843476
Title: Personalized Spine Study Group Registry
Status: Withdrawn | Type: Observational
Why Stopped: Requested by surgeons to pursue new study
Sponsor: Medicrea, USA Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1510
Record Dates: First submitted 2019-02-04; First posted 2019-02-18 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Scoliosis; Adolescence; Degenerative Disc Disease; Spinal Fusion; Kyphoscoliosis; Pseudoarthrosis of Spine; Spinal Stenosis; Kyphoses, Scheuermann
MeSH Terms: conditions — Scoliosis; Intervertebral Disc Degeneration; Spinal Stenosis; Scheuermann Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Surgical with Rod: The patient is being treated with the patient specific rod with a surgery date planned
  Interventions: Device: Patient Specific Rod

INTERVENTIONS:
Device: Patient Specific Rod — Posterior spinal fusion rod
  Other Names: UNiD Rod

SUMMARY:
As a registry, the primary objective of the study is a data collection initiative. The study will collect clinical and radiographic outcomes of patients implanted with Medicrea's PSR. The secondary objective is to collect clinical and radiographic outcomes of patients with Medicrea hardware as a control cohort to the patient-specific rods.

DETAILED DESCRIPTION:
The registry will follow the patient during their standard of care visits. At each visit, the patient will answer questions about themselves and also fill out patient reported outcome sheets. Spinopelvic measurements will be obtained on the x-rays taken. This registry is observational only, and there is no driving hypothesis for data collection. Some broad topics of discussion are:

1. Outcomes of patients sagittal profile through the pre-operative, plan and post-operative events
2. Effectiveness of rod in conjunction with other surgical implants by measurements of fusion assessment and sagittal alignment
3. Outcomes of patients in subgroups as defined by surgery performed, comorbidities, radiographic measurement, or other outcome variables
4. Rod curvature maintenance over the follow-up period
5. Understand the post-operative risks and complications from the pre-operative condition

ELIGIBILITY:
Inclusion Criteria:

* Patient has been/ will be operated and instrumented with PSR from Medicrea
* Patient able to complete a self- administered questionnaires
* Patient able to consent or assent

Exclusion Criteria:

* Patient unable to sign an informed consent form
* Patient unable to complete a self-administered questionnaire
* Patient is pregnant or planning on becoming pregnant during the duration of their study participation
* Patient is older than 85
* Patient is younger than 10

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient is being implanted with patient specific rod
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Data collection initiative | Up to 4 years
  The study will collect clinical and radiographic outcomes of patients implanted with Medicrea's PSR.

SECONDARY OUTCOMES:
Collect clinical and radiographic outcomes of patients with Medicrea hardware | 1 year
  A control cohort to the patient-specific rods

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared with the other investigators in the group